CLINICAL TRIAL: NCT06431737
Title: Comparison of Helicobacter Pylori Eradication Rates Between Twice- and Four-times-daily Amoxicillin Administration in 2-week Tegoprazan-based Triple Therapy: A Propensity Score Matching Analysis
Brief Title: Comparison of Twice- and Four-times-daily Amoxicillin Administration in 2-week Tegoprazan-based H. Pylori Eradication
Status: Completed | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jun-Hyung Cho, Professor, Soonchunhyang University Hospital
Other Study IDs: SCH-HP-2024
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: H.Pylori Infection
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BID group: Tegoprazan 50 mg bid, amoxicillin 1000 mg bid, clarithromycin 500 mg bid for 14 days
  Interventions: Drug: Amoxicillin
- QID group: Tegoprazan 50 mg bid, amoxicillin 500 mg qid, clarithromycin 500 mg bid for 14 days
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — Tegoprazan 50 mg bid, amoxicillin 1000 mg bid or 500 mg qid, clarithromycin 500 mg bid for 14 days

SUMMARY:
Gastric acid depressant play a major role in an H. pylori eradication therapy by (1) increasing the intragastric pH, which improves antibiotic stability and bioavailability; (2) increasing the intragastric pH to 6 or more, which prompts H. pylori to replicate and thus become more sensitive to antibiotics that are effective only against replicating bacteria, such as amoxicillin; (3) increasing the concentration of antibiotics in the stomach. Of antimicrobial agents against H. pylori, amoxicillin is a penicillin derivative that inhibits the synthesis of the bacterial cell wall. Therefore, amoxicillin's bactericidal effect requires the bacteria to be replicating. Amoxicillin is excreted by the kidneys, the plasma half-life is approximately 1 hour, and the bactericidal effect is time dependent. Theoretically, amoxicillin should be given 3 or 4 times daily to maximize the time above minimal inhibitory concentration (MIC) However, in most H. pylori eradication therapies, amoxicillin is given twice daily, where the estimated time above MIC attained by twice daily dosing is insufficient for amoxicillin. Because most strains of H. pylori are sensitive to amoxicillin, 3 or 4 times daily administration may be appropriate to increase the H. pylori eradication success. Nevertheless, data regarding the amoxicillin dosing interval for successful H. pylori eradication are lacking.

DETAILED DESCRIPTION:
The investigators aim to compare the H. pylori eradication rates between twice- and four-times-daily amoxicillin administration in 2-week tegoprazan-based triple therapy. Secondary outcomes are treatment compliance and drug-related adverse event rates.

ELIGIBILITY:
Inclusion Criteria:

* Gastroscopy can be performed
* H. pylori test and pathological analysis can be performed

Exclusion Criteria:

* Age < 20 or > 80 years
* Anemia (serum hemoglobin level < 10 g/dL)
* Severe systemic disease
* Advanced chronic liver disease
* Use of certain medications, including proton pump inhibitors, H2- receptor antagonists, or antibiotics
* History of H. pylori eradication
* Drug allergy to antibiotics
* History of gastric surgery
* Recent history of upper gastrointestinal bleeding

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: H. pylori-infected patients
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
H. pylori eradication rates | 6 weeks
  Urea breath test after completing H. pylori eradication regimen

SECONDARY OUTCOMES:
Treatment compliance | 6 weeks
  Assessment of patients' numbers completing H. pylori eradication regimen
Drug-related adverse event rate | 6 weeks
  Bitter tongue, nausea/vomiting, bloating, diarrhea, and abdominal pain during H. pylori treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Hyung Cho, M.D., Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Soonchunhyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No